CLINICAL TRIAL: NCT03094910
Title: RaynAUT - Thermography and the Autonomic Nervous System in Raynaud's Phenomenon - Investigation of the Autonomic Nervous System in Patients With Raynaud's Phenomenon, Glaucoma, and Autonomic Neuropathy.
Brief Title: Investigation of the Rewarming og the Fingers After Cooling and the Autonomic Nervous System in Raynaud's Phenomenon
Acronym: RaynAUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Lotte Lindberg, Principal investigator, Herlev Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HGH-2016-111; H-16035842 (Other: Research Ethics Committee of the Capital Region)
Record Dates: First submitted 2017-03-08; First posted 2017-03-29 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Raynaud Disease; Raynaud Phenomenon; Hand and Arm Vibration Syndrome; Diabetes Mellitus; Parkinson Disease; Glaucoma; Autonomic Neuropathy; Autonomic Imbalance
Keywords: Raynaud Phenomenon; Hand and Arm Vibration Syndrome; Autonomic Imbalance; Thermography
MeSH Terms: conditions — Raynaud Disease; Hand-Arm Vibration Syndrome; Diabetes Mellitus; Parkinson Disease; Glaucoma | interventions — Tilt-Table Test; Thermography; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 123I-MIBG (Other): Only the group of participants with primary Raynaud's phenomenon (Raynaud's disease) is also scheduled for this intervention, the 123I-MIBG.
  Interventions: Diagnostic Test: Examination of vibration perception threshold in fingertips; Diagnostic Test: Ewing's tests; Diagnostic Test: Tilt table test; Diagnostic Test: Thermography; Diagnostic Test: 123I-MIBG; Diagnostic Test: Blood samples
- All participants (Other): Examination of vibration perception threshold in fingertips, thermography, Ewing's test, tilt table test, blood samples.
  Interventions: Diagnostic Test: Examination of vibration perception threshold in fingertips; Diagnostic Test: Ewing's tests; Diagnostic Test: Tilt table test; Diagnostic Test: Thermography; Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Examination of vibration perception threshold in fingertips — Vibration perception threshold is examined for 7 different frequences. All fingers are examined except for the thumbs.
Diagnostic Test: Ewing's tests — A battery of tests invented to diagnose the cardiac autonomic neuropathy in diabetics. Heart rate and blood pressure are measured during Valsalva maneuver, deep breathing, active standing and prolonged handgrip.
Diagnostic Test: Tilt table test — Blood pressure and heart rate are measured continuously while the participant is brought to a 60 degree position and held there for 15 minutes.
Diagnostic Test: Thermography — An infrared thermographic camera is applied to record temperature of the fingers of the participant before and after cooling in 10 degree water for 1 min.
Diagnostic Test: 123I-MIBG — 123I-MIBG is injected into a vein, and an early and a late scan is performed. Regions Of Interest are selected for the heart and mediastinum, and the ratio as well as well as the Washout Rate can be determined. MIBG is a noradrenaline analogue and the examination is performed to visualize a potential imbalance of the autonomic nervous system of the heart.
  Arms: 123I-MIBG
Diagnostic Test: Blood samples — The blood samples will be assayed for hemoglobin, long-term blood sugar, C-reactive protein, sodium, potassium, magnesium, albumin, TSH, vitamin B and D, and ionized calcium.
  Patients with suspected Raynaud's disease will be tested for anti-nuclear antibodies (ANA) to screen for underlying rheumatic illness.
  Blood samples will also be drawn during tilt table testing and assayed for plasma catecholamines.

SUMMARY:
Patients with Raynaud's disease have an increased tendency of chest pain and migraine, and studies indicate that the disease might be associated with increased cardiovascular morbidity and mortality. Furthermore, a certain hyperactivity of the sympathetic nervous system has been demonstrated in these patients. Hyperactivity of the sympathetic nervous system is known to cause decreasing heart function, regardless of the underlying disease.

The cardiac autonomic nervous function and thermographic parameters will be assessed in patients with primary and secondary Raynaud's phenomenon and glaucoma as well as in patients diagnosed with autonomic dysfunction such as diabetics and patients with Parkinson's disease in order to compare the function of the cardiac autonomic nervous system and the peripheral response to cold exposure. Potentially, this will lead to a better understanding of the cardiac autonomic nervous function in Raynaud's phenomenon. Moreover, it might give rise to a new perception of the condition and its association to cardiovascular disease.

At the Department of Clinical Physiology, the current method of detecting Raynaud's phenomenon is time-consuming and unpleasant to the patient due to cooling for several minutes. Another aim of the PhD study is to implement infrared thermography as a gentler and possibly more sensitive method to replace the currently applied method.

The project will also include an epidemiological study based on data obtained from the National Patient Registry, among others. Raynaud's phenomenon will be paired with diagnostic codes of conditions such as diabetes mellitus, Parkinson's disease, glaucoma, and cardiovascular disease.

DETAILED DESCRIPTION:
Raynaud's phenomenon:

Raynaud's phenomenon is defined by vasospasms occurring in the fingers, toes, nose, ears or tongue lasting for minutes to hours. The attacks of vasospasms are provoked by cold exposure or stressful emotions and present themselves as well demarcated pallor of the skin and may include desensitization of the discolored area. Then cyanosis and eventually redness occur due to post ischemic hyperemia, which also can give rise to paresthesia and pain.

The phenomenon can be divided into a primary, idiopathic form - Raynaud's disease - that represents up to 90 % of all cases of Raynaud's phenomenon, is seen primarily in patients less than 40 years, and is usually considered benign. While the secondary form is often associated with rheumatic disorders such as scleroderma, it is also seen connected to other diseases, including vibration injury, external compression (e.g. a neck rib), medication, and vascular disorders such as atherosclerosis.

The prevalence of Raynaud's phenomenon varies among studies according to diagnostic criteria and geography as the climate affects the occurrence: In Northern Europe 15-20 % of the population is affected while the prevalence is 2-5 % in Southern Europe. An increased prevalence of migraine, chest pain, including Prinzmetal's angina, has been demonstrated in patients with Raynaud's disease. A study with 3,442 participants found an association between Raynaud's disease and cardiovascular disease, including ischemic heart disease, intermittent claudication, heart failure and cerebrovascular disease. Furthermore, an increased mortality has been found in Caucasian patients with Raynaud's disease. Consequently, Raynaud's disease might be a sign of or a precursor to cardiovascular disease.

Documentation of Raynaud's phenomenon:

Infrared thermography is a method of detecting infrared energy and converting it into a video signal. The method is non-invasive; in fact the method requires no contact between the camera and the investigated object. Previously, the method has been compared to reference methods for demonstrating Raynaud's phenomenon and has been evaluated in extensive reviews. Infrared thermography is a gentler and potentially more sensitive method of demonstrating Raynaud's phenomenon. It may replace the method of systolic blood pressure with cold provocation resulting in a less unpleasant examination to the patient.

The nervous system:

The exact mechanism of Raynaud's phenomenon is yet to be clarified. However, the sympathetic nervous system plays an important role in the process. A lack of habituation of the sympathetic response to a sound stimulus has been demonstrated in patients with Raynaud's disease compared to healthy participants who demonstrated normal habituation. Furthermore, a sensitization of the physiologic response to cold has been proposed, advocating an altered central control of the peripheral nervous system. A certain hyperactivity of the sympathetic nervous system has been demonstrated in patients with Raynaud's disease, supporting the theory that an autonomic abnormality might accompany Raynaud's disease.

123I-MIBG scintigraphy: The cardiac sympathetic activity can be visualized by a radio tracer, the norepinephrine-analogue metaiodobenzylguanidine (MIBG) marked with Iodine-123. An increased activity of the sympathetic nervous system is visualized by a decreased late heart/mediastinum ratio and an increased washout rate. This method is not widely applied in the clinical setting, and it is primarily employed in research projects involving patients with heart failure whose sympathetic nervous system is chronically hyperactive leading to progression of heart failure. However, it has been demonstrated that the method is also able to visualize abnormal sympathetic nervous activity in patients with preserved ejection fraction, to distinguish reversible and irreversible cardiac autonomic neuropathy in diabetics [15;16], and to act as a sensitive marker of autonomic dysfunction in patients with Parkinson's disease.

Autonomic dysfunction:

Diabetes Mellitus and Parkinson's disease often give rise to autonomic dysfunction. Cardiac autonomic neuropathy (CAN) is a type of abnormal autonomic nervous function that precipitates abnormal heart frequency and blood pressure. CAN is present in approximately 20 % of diabetics. In the 1970s, David Ewing developed various tests to demonstrate autonomic dysfunction in diabetics. The relation between the sympathetic and the parasympathetic nervous system can be further demonstrated by analyzing the heart rate variability (HRV) during rest. This is a simple measure of altered cardiac autonomic control and seems to be a good predictor of cardiovascular disease. Initially, CAN causes an increased heart frequency due to decreased parasympathetic activity. Subsequently, sympathetic tone decreases; the heart frequency decreases accordingly and remains stable without its normal variability. With further progression CAN leads to increased cardiovascular morbidity and mortality.

Glaucoma:

The relationship between normal-pressure glaucoma and autonomic dysfunction measured by perimetry and heart rate variability, respectively, was evaluated in a study where parasympathetic activity was found to be decreased, and the sympathetic activity as well as the interrelating ratio increased in patients with normal-pressure glaucoma compared to healthy age-matched participants. These findings indicate that the sympathetic activity in patients with normal-pressure glaucoma is raised above normal.

Purpose of the project:

The overall purpose of the project is to elucidate the peripheral and the central parts of the autonomic nervous system and to demonstrate their contribution to different diseases - diseases that are generally perceived as either peripheral or central in origin.

The investigation will be done by means of thermography, tilt table test, blood samples, physiological tests, scintigraphy of the heart, and test of tactile sensitivity.

For example, in Raynaud's disease the vasospasms of the fingers or toes are the main feature. However, in the literature there seems to be an association between these peripheral attacks and vasospasms in other organs such as the heart and the brain, assumingly causing Prinzmetal's angina and migraine, respectively. Furthermore, a certain hyperactivity of the sympathetic nervous system in Raynaud's disease has been reported in the literature and should be further studied.

While 123I-MIBG has been demonstrated to be able to detect sympathetic hyperactivity in various patients, supposedly, 123I-MIBG has never been performed in patients with Raynaud's disease. Abnormal findings applying this method as well as the autonomic tests of Ewing in these patients would be a strong indication of a general imbalance of the cardiac autonomic nervous system.

Ultimately, it will question the general perception that Raynaud's disease is a harmless condition. An association with autonomic dysfunction could be the link between Raynaud's disease and the increased cardiovascular morbidity and mortality suggested in these patients in the literature.

Objectives:

The overall objectives of the project is partly to implement the method of infrared thermography as a new method of detecting Raynaud's phenomenon, and partly to investigate whether Raynaud's disease is part of a generalized autonomic neuropathy giving rise to not only peripheral vasospasms. During the project, the cardiac autonomic nervous system will be investigated in patients with Raynaud's phenomenon, in patients diagnosed with autonomic dysfunction as well as in patients with normal-pressure glaucoma as they similarly to patients with Raynaud's disease supposedly have an increased sympathetic activity.

Additionally, the project will include an epidemiologic study based on data obtained from e.g. the National Patient Registry where Raynaud's phenomenon is paired with conditions such as diabetes mellitus, Parkinson's disease, glaucoma, and cardiovascular disease in an attempt to estimate their respective relationship to Raynaud's phenomenon.

Subjects and methods:

Participants:

The project will involve the following groups of participants:

1. Patients with primary Raynaud's phenomenon/Raynaud's disease
2. Patients with secondary Raynaud's phenomenon, primarily vibration-induced
3. Patients suspected of having Raynaud's phenomenon, referred for examination
4. Patients with diabetes mellitus
5. Patients with Parkinson's disease
6. Patients with normal-pressure glaucoma
7. Healthy participants, preferably age- and gender-matched with the respective groups of patients

To be able to obtain statistical power, 20 patients will be included in each of the groups 1-6. Some of the groups are dominated by a certain gender and/or age range. Accordingly, 40 participants will be recruited to the group of healthy participants (group 7) to be able to match the other groups by age and gender.

Examinations:

The project consists of various examinations as described below. Infrared thermography, physiological examinations, sensitivity test, and blood samples will be performed on all groups of participants. In addition, 123I-MIBG will be performed on patients with Raynaud's disease only.

1. Infrared Thermography This method should be able to detect Raynaud's phenomenon by recording the ability of the fingers to recover baseline temperature after cooling.

   Initially, the baseline temperature of the hands is recorded by taking a thermographic picture. The participant's hands are immersed in cold water (10 °C) for 1 minute, and the infrared camera records the temperature recovery in a video sequence.

   The temperature recovery will be analyzed by at least 10 different variables (curve analysis and visual inspection).
2. Physiological examinations All patients will be examined applying

   - Ewing's tests: Deep breathing, Valsalva maneuver, active standing, and sustained handgrip. During the tests, heart rate and blood pressure will be measured continuously.
   * Five minutes of resting during continuous measurements of heart rate and blood pressure.
   * Tilt table test After resting in a supine position the patient is tilted to 60° for 15 minutes during which heart rate and blood pressure are measured continuously. Blood samples are drawn before and after the tilt in order to analyze the hormonal stress response.
3. Sensitivity test Sensitivity to vibration in the fingers is examined using the Vibrosense Meter®. Vibration with seven different frequencies is applied to the fingers, each with alternating intensity, and the threshold for vibration for each patient can be assessed as the participant removes his/her finger from a button when vibration is no longer perceptible.
4. Blood samples On the day of the examinations the blood samples will be drawn via the Department of Clinical Biochemistry. These blood tests are intended to rule out possible differential diagnoses to abnormal physiological or sensitivity tests. The blood samples will be assayed for hemoglobin, long-term blood sugar, C-reactive protein, sodium, potassium, magnesium, albumin, TSH, vitamin B and D, and ionized calcium. Patients with suspected Raynaud's disease will be tested for anti-nuclear antibodies (ANA) to screen for underlying rheumatic illness.

   Blood samples will also be drawn during tilt table testing and assayed for plasma catecholamines. At the same time, a sample of plasma and serum will be drawn for possible future analysis. A research biobank is created for this purpose.
5. 123I-MIBG 123I-MIBG scintigraphy will be performed on patients with Raynaud's disease to visualize whether the cardiac sympathetic nervous system is in fact affected by this disease.

ELIGIBILITY:
Criteria depend on the specific group of participants. Criteria described below are applicable to the group of participants with Raynaud's syndrome

Inclusion Criteria:

- Attacks of demarcated pallor of the skin of the fingers provoked by exposure to cold

Exclusion Criteria:

* Positive Anti-Nuclear Antibodies
* Connective tissue disease
* Current smoker
* Current treatment with beta blocker
* Other predisposing factors for developing Raynaud's phenomenon
* Pacemaker
* Cardiac arrhythmia
* Pregnancy
* Diabetes mellitus
* Parkinson's disease
* Glaucoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Thermography of the hands after cooling - a composite evaluation of the rewarming ability | Participant is examined once for a maximum of 1 hour.
  Determination of which variables are able to distinguish the participants with Raynaud's phenomenon from the healthy participants.
  Temperature (degrees celsius), time (minutes), degrees/min, acceleration of temperature change (degrees/min^2), recovery index (percent).
  All measurements will be evaluated in terms of ability to diagnose Raynaud's phenomenon. Finally, the most prominent variables are aggregated to determine whether or not the participant has Raynaud's phenomenon or not.
Heart rate variability (HRV) | Participant is examined once for 1,5 hours.
  Determination of HRV from participants with Raynaud's phenomenon, with diagnosed autonomic neuropathy, and healthy participants. All measurements will be aggregated to determine whether HRV differs among the different groups of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lars T Jensen, DMSc, Study Director — Department of Clinical Physiology, Herlev Hospital
Locations (1):
- Department of Clinical Physiology and Nuclear Medicine, Herlev Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindberg L, Kristensen B, Thomsen JF, Eldrup E, Jensen LT. Characteristic Features of Infrared Thermographic Imaging in Primary Raynaud's Phenomenon. Diagnostics (Basel). 2021 Mar 20;11(3):558. doi: 10.3390/diagnostics11030558. PMID 33804657